CLINICAL TRIAL: NCT04476901
Title: A Phase IIB Randomized, Placebo-Controlled, Multicenter Study of the Comparative Efficacy and Safety of Administration of Allogeneic-MSC Versus Placebo in Patients With Non- Ischemic Dilated Cardiomyopathy
Brief Title: Administration of Allogeneic-MSC in Patients With Non-Ischemic Dilated Cardiomyopathy
Acronym: DCMII
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joshua M Hare (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Principal Investigator, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200566; CDMRP-PR191597 (Other Grant/Funding Number: US Department of Defense); 20-02-134 (Other: BRANY IRB)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Non-ischemic Dilated Cardiomyopathy
Keywords: Allogeneic mesenchymal stem cells; Bone marrow-derived mesenchymal stem cells

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Genotype A administered with placebo Group (Placebo Comparator): Participants whose blood genotyping resulted with Genotype A (absence of any variant/ presence of benign variant) and randomized to the placebo group will receive the placebo intervention.
  Interventions: Other: Placebo
- Genotype A administered with hMSC Group (Experimental): Participants whose blood genotyping resulted with Genotype A (absence of any variant/ presence of benign variant) and randomized to the treatment group will receive the hMSC intervention.
  Interventions: Biological: allogeneic human mesenchymal stem cells (hMSCs)
- Genotype B administered with placebo Group (Placebo Comparator): Participants whose blood genotyping resulted with Genotype B (variants of uncertain significance) and randomized to the placebo group will receive the placebo intervention.
  Interventions: Other: Placebo
- Genotype B administered with hMSC Group (Experimental): Participants whose blood genotyping resulted with Genotype B (variants of uncertain significance) and randomized to the treatment group will receive the hMSC intervention.
  Interventions: Biological: allogeneic human mesenchymal stem cells (hMSCs)
- Genotype C administered with placebo Group (Placebo Comparator): Participants whose blood genotyping resulted with Genotype C (pathogenic or likely pathogenic variants) and randomized to the placebo group will receive the placebo intervention.
  Interventions: Other: Placebo
- Genotype C administered with hMSC Group (Experimental): Participants whose blood genotyping resulted with Genotype C (pathogenic or likely pathogenic variants) and randomized to the treatment group will receive the hMSC intervention.
  Interventions: Biological: allogeneic human mesenchymal stem cells (hMSCs)

INTERVENTIONS:
Biological: allogeneic human mesenchymal stem cells (hMSCs) — allo-hMSCs, 16-20 million cells/ml delivered at a dose of 0.5 ml/ injection x 10 injections for a total of 80-100 million allo-hMSCs or a single administration of intravenous allogeneic hMSCs (100 million).
  Arms: Genotype A administered with hMSC Group; Genotype B administered with hMSC Group; Genotype C administered with hMSC Group
Other: Placebo — Placebo will be administered as injections of plasmalyte A supplemented with 1% of 25% human serum albumin (HSA). 0.5 ml/ injection x 10 injections or an intravenous placebo infusion of Cell-free PlasmaLyte-A medium supplemented with 1% of 25% human serum albumin (HSA)
  Arms: Genotype A administered with placebo Group; Genotype B administered with placebo Group; Genotype C administered with placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an experimental drug called human allogeneic mesenchymal stem cell therapy.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Men and women aged 18 to 80 years (inclusive) at the time of signing the informed consent form.
2. Diagnosis of NIDCM with left ventricular ejection fraction ≤45%.
3. Appropriate guideline-directed optimal medical therapy for non-ischemic cardiomyopathy. At a minimum, subjects must be on beta blockers and angiotensin-converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs) or Angiotensin Receptor Neprilysin Inhibitors (ARNI) or have appropriate medical indication precluding use of one or both of these agents. Subjects must be on a stable regimen for at least 30 days prior to the procedure. Dose titration is allowed.
4. Be a candidate for cardiac catheterization*
5. Be willing to undergo DNA test.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Be eligible for or require standard-of-care surgical or percutaneous intervention for the treatment of non-ischemic dilated cardiomyopathy
2. Clinical manifestation of coronary artery disease (CAD) (e.g., chest pain and concomitant clinical findings such as electrocardiogram changes suggestive of coronary ischemia, myocardial infarction) or evidence of endocardial or transmural scar on cardiac MRI suggestive of undiagnosed CAD or history of percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG). Be indicated for or require coronary artery revascularization
3. Documented presence of epicardial stenosis of 70% or greater in one or more major epicardial coronary arteries
4. Valvular heart disease including 1) aortic valve prosthesis, mechanical mitral valve, and mitral valve clip; 2) severe aortic valve insufficiency/regurgitation within 12 months of consent*
5. Aortic stenosis with valve area ≤ 1.5cm2*
6. Cardiomyopathy due to acute Post-partum (within 6 months), Non-compaction*, or Hypertrophic* cardiomyopathy
7. Cardiomyopathy due to known toxin (e.g amyloid) Note: anthracycline induced cardiomyopathy will be allowed
8. QTc interval > 550 ms on baseline electrocardiogram (ECG) (note: QTc interval is the interval between the start of the Q wave and the end of the T wave in the heart's electrical cycle)
9. Automated Implantable Cardioverter Defibrillator (AICD) appropriate firing or anti tachycardia pacing for ventricular tachycardia or ventricular fibrillation within 30 days prior to consent
10. Have an estimated baseline glomerular filtration rate below the clinical site's institutional cutoff
11. A hematologic abnormality during baseline testing as evidenced by hemoglobin < 9 g/dl; hematocrit < 30%; absolute neutrophil count < 2,000 or total WBC count more than 2 times upper limit of normal; or platelet values < 100,000/ul
12. Have liver dysfunction, as evidenced by enzymes Aspartate Transaminase Enzyme (AST) and Alanine Aminotransferase Enzyme (ALT) greater than three times the ULN
13. Have a bleeding diathesis or coagulopathy (International Normalised Ratio (INR) > 1.5), cannot be withdrawn from anticoagulation therapy, or will refuse blood transfusions
14. Be a solid organ transplant recipient. This does not include prior cell based therapy (>12 months prior to enrollment), bone, skin, ligament, tendon or corneal grafting.
15. Have a history of organ or cell transplant rejection
16. Have a clinical history of malignancy within the past 12 months (i.e., subjects with prior malignancy must be disease free for 12 months), except curatively treated basal cell or squamous cell carcinoma or cervical carcinoma
17. Drug and/or alcohol abuse or dependence within the past 9 months
18. Be serum positive for HIV, hepatitis B surface antigen, or viremic hepatitis C
19. Documented presence of a known Left Ventricular (LV) thrombus, aortic dissection, or aortic aneurysm. (Refer to "Guidance to the PI" section with regards to LV thrombus, below)*
20. Blood glucose levels (HbA1c) >10%
21. Severe radiographic contrast allergy
22. Known history of anaphylactic reaction to penicillin or streptomycin
23. Hypersensitivity to dimethyl sulfoxide (DMSO)
24. Non-cardiac condition with life expectancy < 1 year
25. Acute stroke or transient ischemic attack within 3 months of enrollment
26. Be pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods
27. Pacemaker-dependence with an Implantable Cardioverter Defibrillator (ICD) (Note: pacemaker-dependent candidates without an ICD are not excluded)
28. Presence of a pacemaker and/or ICD generator with any of the following limitations/conditions:

    * manufactured before the year 2000
    * leads implanted < 6 weeks prior to consent
    * non-transvenous epicardial or abandoned leads
    * subcutaneous ICDs
    * leadless pacemakers
29. A cardiac resynchronization therapy (CRT) device implanted less than 3 months prior to consent
30. Other MRI contraindications (e.g. subject body habitus incompatible with MRI)
31. Need for advanced heart failure therapy (e.g. IV inotropes)
32. Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial
33. Any other condition that in the judgment of the Investigator would be a contraindication to enrollment or follow-up

(*) Applies to subjects receiving product via transendocardial administration only

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in LVEF | Baseline, 12 months
  Change in Left Ventricular Ejection Fraction (LVEF) as assessed via cardiac Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Change in global ventricular strain | Baseline, 12 months
  Change in global ventricular strain as assessed via cardiac Harmonic Phase (HARP) MRI
Change in left regional strain | Baseline, 12 months
  Change in regional ventricular strain as assessed via cardiac HARP MRI
Left ventricular function concordance | 12 months
  The left ventricular function concordance will be measured as the Number of individuals who experienced an increase in left ventricular ejection fraction (LVEF) and a simultaneous decrease in both left ventricular end systolic volume index (LVESVI) and left ventricular end diastolic volume index (LVEDVI)
Change in LVEDVI | Baseline, 12 months
  Change in left ventricular end diastolic index (LVEDVI) as assessed via cardiac MRI
Change in LVESVI | Baseline, 12 months
  Change in left ventricular end systolic index (LVESVI) as assessed via cardiac MRI
Change in Maximal oxygen consumption (peak VO2) | Baseline, 12 months
  Change in maximal oxygen consumption (peak VO2) as assessed via treadmill
Change in Exercise tolerance | Baseline, 12 months
  Change in exercise tolerance as assessed as the distance covered via the six-minute walk test
Change in Minnesota Living with Heart Failure Questionnaire (MLHFQ) Score | Baseline, 12 months
  Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a 21-item questionnaire with a total score ranging from 0 to 105 with lower scores indicative of better outcome.
Change in New York Heart Association (NYHA) Class | Baseline, 12 months
  NYHA Classifications of heart failure are as follows: Class I (no limitations); Class II (mild symptoms); Class III (marked limitations); Class IV (Severe limitations)
Percent change in flow mediated diameter | Baseline, 12 months
  Change in endothelial function will be reported as the percent change in flow mediated diameter assessed via flow mediated dilation (FMD).
Change in EPC-CFU | Baseline, 12 months
  Change in endothelial function will be reported as the change in Endothelial Progenitor Cell Colony Forming Unit (EPC-CFU) assessed via blood sample assay
Change in N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) | Baseline, 12 months
  Change in NT-proBNP as assessed via blooddraw
Change in cytokines | Baseline, 12 months
  Change in NT-proBNP as assessed via blooddraw
Incidence of MACE | 12 months
  Safety will be reported as the incidence of Major Adverse Cardiac Events (MACE) assessed by treating physician
Incidence of TE-SAEs | Day 30
  Safety will be reported as the incidence of Treatment Emergent Serious Adverse Events (TE-SAEs) assessed by treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hare, MD, Principal Investigator — University of Miami
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Louisville, Louisville, Kentucky
  - Texas Heart Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cardiovascular Cell Therapy Research Network — https://www.cctrn.org
- See also: Information on stem cells from the National Institutes of Health — https://stemcells.nih.gov/
- See also: DCM II Trial — https://www.dcmii.org